CLINICAL TRIAL: NCT00936039
Title: The Effect of Immobilization on Myocellular Characteristics in Healthy, Young Males
Brief Title: Effects of Unloading on Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEC-09-3-011
Record Dates: First submitted 2009-07-06; First posted 2009-07-09 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Immobilization; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unloading (Experimental): 2 weeks of unloading
  Interventions: Behavioral: unloading

INTERVENTIONS:
Behavioral: unloading — 2 weeks of unloading of a single leg

SUMMARY:
In the present study, the effects of 3 weeks of unloading on muscle mass and muscle fiber characteristics will be determined. In addition, the effects of 6 weeks of recovery will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI < 30 kg/m2

Exclusion Criteria:

* Use of medication that may affect haemostasis
* Subjects with (recent) musculoskeletal/orthopaedic disorders known to affect the outcome of the study or that compromise their ability to walk with crutches
* Subjects with metal implants in their lower limbs
* Subjects with known cardiovascular and/or haemostasis disorders
* Subjects with known severe hypertension

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
muscle mass, muscle fiber size | 1 week before unloading; immediately (1 day) after unloading and 6 weeks after unloading

SECONDARY OUTCOMES:
muscle strength | 1 week before unloading; immediately (1 day) after unloading and 6 weeks after unloading

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356